CLINICAL TRIAL: NCT06269159
Title: The Power of 24-hour: Co-designing Intervention Components to Stimulate 24-hour Movement Behaviors in Adults With Overweight and Obesity
Brief Title: The Power of 24-hour: Co-designing Intervention Components
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0185
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Overweight and Obesity
Keywords: Concept mapping; physical activity; sedentary behavior; qualitative research
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care providers: 10 health care providers: physiotherapist working with adults with overweight and obesity
  Interventions: Other: Concept mapping: brainstorm; Other: Concept mapping: clustering and rating
- Adults with overweight and obesity: Inclusion criteria
  * Adults aged 25-64 years
  * Active on the job market for at least 50 percent
  * BMI ≥25kg/m²
  Exclusion criteria
  * Retirement and early retirement
  * Unemployment
  * Working for less than 50 percent
  * Working in night shifts
  * Physical (e.g. amputations, paralysis, recovering from stroke, osteoarthritis), cognitive (e.g. dementia, psychological disorders) and major medical (e.g. Chronic respiratory diseases, heart failure, cardiovascular diseases, cancer) conditions that obstruct daily functioning
  * Diabetes diagnosed by a general practitioner
  * Pregnancy
  * Pregnancy <1 year ago
  * Currently involved in study specific weight loss interventions
  * Post-surgery weight loss interventions
  * Waitlist for weight loss surgery
  * Hospitalized
  Interventions: Other: Concept mapping: brainstorm; Other: Concept mapping: clustering and rating

INTERVENTIONS:
Other: Concept mapping: brainstorm — Group health care providers:
  * Duration: 1.5 hour for HCP via zoom session
  * Brainstorm question: what would help your clients to change their sedentary behavior into more physical activity?
  Group adults with overweight and obesity
  * Duration: online survey (REDCAP) of approx. 10 minutes
  * Brainstorm question via an online survey. What would help you to change your sedentary behavior into more physical activity?
Other: Concept mapping: clustering and rating — The same participant of the brainstorm session are asked to join session 2 to complete the clustering and rating). All interested adults will get access to the online cluster and rate tool described below.
  * Duration: flexible use of the online tool (available for two weeks)
  * The clustering and rating of all needs mentioned in session 1 will be done online and individually via a web application. In this online tool, the final list of 'needs' generated in session 1 will be presented.
  * Individually sort the 'needs' into groups and give the group a theme. In addition, each need will be scored on effectiviness, feasibility, modifiability. Thhe participants have unlimited access for two weeks.

SUMMARY:
Most of the existing lifestyle interventions in adults with overweight or obesity focus on one movement behavior in isolation (i.e. moderate to vigorous physical activity (MVPA)). However, recent research suggests to incorporate all movement behaviors performed in one day to explore the possible synergistic health effects of targeting more than one behavior. Moreover, more optimal 24-hour movement behavior compositions are related with better cardiometabolic health. Literature shows that adults with obesity have less optimal 24-hour compositions (8-9). Therefore it would be of interest to discover the needs related to an optimal 24-hour movement behavior intervention for a group of adults with overweight and obesity using co-design to develop an intervention.

This study will conduct a concept mapping protocol to explore the needs to of people with overweight and obesity to change their sedentary behavior into more physical activity as well to include the opinion of health care providers (HCP are physiotherapists) on the needs of their patients.

ELIGIBILITY:
Group Health Care providers

Inclusion Criteria:

* The HCP will consist of physiotherapists and movement on referral coaches (https://www.gezondleven.be/projecten/bewegen-op-verwijzing). HCP are included when working on a healthy lifestyle as well as working with clients struggling with overweight or obesity.

Group Adults with overweight and obesity

Inclusion Criteria:

* Adults aged 25-64 years
* Active on the job market for at least 50 percent
* BMI ≥25kg/m²

Exclusion Criteria:

* - Retirement and early retirement
* Unemployment
* Working for less than 50 percent
* Working in night shifts
* Physical (e.g. amputations, paralysis, recovering from stroke, osteoarthritis), cognitive (e.g. dementia, psychological disorders) and major medical (e.g. Chronic respiratory diseases, heart failure, cardiovascular diseases, cancer) conditions that obstruct daily functioning
* Diabetes diagnosed by a general practitioner
* Pregnancy
* Pregnancy <1 year ago
* Currently involved in study specific weight loss interventions
* Post-surgery weight loss interventions
* Waitlist for weight loss surgery
* Hospitalized

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of health care providers as a group of adults with overweight and obesity will be included.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Themes | After session 2 clustering and rating
  Themes will be created that bundle different factors explaining needs to change sedentary behavior into more physical activity for both the group of health care providers as the group of adults with overweight and obesity
Score of effectiveness | After session 2 clustering and rating
  Each need will be scored on effectiveness by both the health care providers as the groups adults with overweight and obesity.
  How effective do you think the 'need' is. Likert scale of 1-5.
Score of feasibility | After session 2 clustering and rating
  Each need will be scored on feasibility by both the health care providers as the groups adults with overweight and obesity. How feasible do you think the 'need' is. Likert scale of 1-5.
Score of modifiability | After session 2 clustering and rating
  Each need will be scored on modifiability by both the health care providers as the groups adults with overweight and obesity. How modifiable do you think the 'need' is. Likert scale of 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lapauw, Principal Investigator — University Hospital, Ghent; Marieke De Craemer, Principal Investigator — University Ghent
Locations (1):
- Ghent university Hospital, Ghent, Belgium